CLINICAL TRIAL: NCT06836687
Title: Monocentric Study to Investigate the Effect of the New Definition of Epilepsies of the International League Against Epilepsy of 2014 on the Diagnosis After the First Seizure, on Patient Satisfaction, Cognition and Health Economic Factors
Brief Title: Effect of the New Definition of Epilepsies of the ILAE of 2014 on the Diagnosis After the First Seizure
Acronym: EFS-ILAE2014
Status: Recruiting | Type: Observational
Sponsor: University Hospital Marburg (Other)
Responsible Party: Principal Investigator, Lena Habermehl, Dr. med., attending staff, University Hospital Marburg
Other Study IDs: AZ 199/17
Record Dates: First submitted 2024-03-19; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Seizure, Epileptic; Neuropsychology; Outcome
Keywords: First epileptic seizure; Definition of epilepsy; Neuropsychology; outcome
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The present study is a prospective study on the development of seizure frequency, medication adherence, quality of life and cognitive performance after a first epileptic seizure using the new diagnostic criteria for epilepsy of the International League Against Epilepsy of 2014 at the time of diagnosis.

DETAILED DESCRIPTION:
The new diagnostic criteria for epilepsy, which have been in place since 2014, suggest that due to the improved possibilities for early diagnosis and treatment - particularly as a result of improved imaging diagnostics - changes in the incidence rates and severity of the course of epilepsies with different etiologies can be expected.

The group of epilepsies with unclear etiology should now be smaller than in previous studies. The MRI- and EEG-positive patients can now be identified as having structural epilepsy based on the type of lesion, which was not possible in previous studies without differentiated imaging. The fact that these patients can now be treated before a patients can now be treated before a second seizure, the risk of recurrence and the health economic costs should also be reduced and have a positive effect on maintaining cognitive performance and quality of life after a first epileptic seizure.

The aim of the study is to record the consequences of the new epilepsy diagnostic criteria in terms of outcome and treatment. In addition, the investigators will use a questionnaire battery and neuropsychological testing to record the potential neuropsychological deficits, financial and socio-medical consequences of a first seizure or early-stage epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the 18th year of life
* first epileptic seizure
* Ability to understand the patient information and to give written consent
* Written consent for voluntary participation in the study

Exclusion Criteria:

* Chronic drug or alcohol abuse in the last two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with an nunprovoked epileptic seizure
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2038-04-01 (Estimated); Study Completion 2038-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of seizure recurrency | 10 Years
  Seizure recurrency is recorded 6 months, 1 year, 3 years, 5 years and 10 years after the first seizure

SECONDARY OUTCOMES:
employment | 10 years
  Currently working as employee or independent, retirement or long-time sick-leave at the first attack, after 6 months, 1, 3, 5 and 10 years.
Salary | 10 years
  Gross salary in Euro at the first attack, after 6 months, 1, 3, 5 and 10 years.
Driving restriction | 10 Years
  Fitness to drive (yes/no) is assessed after the first attack, after 6 months, 1, 3, 5 and 10 years.
Verbale Lern- und Merkfähigkeitstest | 10 years
  Verbale Lern- und Merkfähigkeitstest - VLMT (Helmstaedter, Lendt, & Lux, 2001) at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  0 to 135 points, O worst, 135 best possible result.
Regensburger Wortflüssigkeits-Test | 10 Years
  Regensburger Wortflüssigkeits-Test - RWT (Aschenbrenner, Tucha, & Lange, 2000) at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  Number of words starting with one asked letter, that can be said in 2 minutes (typically between 0 and 50)
Copy and recall of the Rey-Osterrieth Figure | 10 Years
  Copy and recall of the Rey-Osterrieth Figure (Berry, Allen, & Schmitt, 1991) at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  0 to 36 points. 0 worst possible result, 36 best possible result.
Trailmaking Test A & B | 10 Years
  Trailmaking Test A & B (Tombaugh, 2004) at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  individual time to absolve the test in seconds
Wechsler Adult Intelligence Scale - WAIS IV | 10 Years
  Wechsler Adult Intelligence Scale - WAIS IV at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  Intelligence quotient (40 to 160)
TAP | 10 Years
  Test for Attentional Performance - TAP (Zimmermann & Fimm, 2002) at baseline and then after 1 years, 5 years and 10 years after the first seizure:
  reaction time in ms, standard deviation of the reaction time, ratio of errors ratio of correct reactions
Relationsship status | 10 years
  Relationship status (single, maried, divorced) is assessed after the first attack, after 6 months, 1, 3, 5 and 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- c/o Klinik für Neurologie, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weil J, Linka L, Gurschi M, Kidik SA, Fuchs A, Schoenfeldt R, Zahnert F, Moller L, Menzler K, Kemmling A, Knake S, Habermehl L. The impact of white matter lesions on seizure recurrence after first epileptic seizures in the elderly: a prospective study. Neurol Res Pract. 2025 May 20;7(1):36. doi: 10.1186/s42466-025-00391-2. PMID 40394715